CLINICAL TRIAL: NCT03362853
Title: A Randomized, Single-center, Placebo and Positive Control, 4-period and 4-crossover Clinical Study Evaluating the Effect of a Single-dose Oral Administration of Nemonoxacin Malate Capsule on QTc Intervals and Heart Rhythms of Healthy Subjects as Well as the Influence of Food Intake on QTc Intervals and Pharmacokinetic Characteristics
Brief Title: A Study Evaluating the Effect of a Single-dose Oral Administration of Nemonoxacin Capsule on QTc Intervals and Heart Rhythms of Healthy Subjects and the Influence of Food Intake on QTc Intervals and Pharmacokinetic Characteristics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TaiGen Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TG-873870-C-7
Record Dates: First submitted 2017-11-23; First posted 2017-12-05 (Actual); Last update posted 2017-12-06 (Actual); Status verified 2017-12

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — nemonoxacin; Moxifloxacin; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Stage I: the administration sequences of the 4 groups were CABD, ADCB, BCDA and DBAC respectively. D represents moxifloxacin, the positive control drug, for which an open design was adopted. For the other 3 groups, i.e. 500 mg nemonoxacin, 750 mg nemonoxacin, and placebo, a double-blind design was employed.
  Stage II: An open design for 12 subjects who had completed Stage I to receive a single oral dose of 500 mg nemonoxacin after taking a high-fat test meal
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Nemonoxacin 500Mg Capsule (Experimental)
  Interventions: Drug: Nemonoxacin 500Mg Capsule; Drug: Moxifloxacin 400Mg Tablet; Drug: Nemonoxacin 750Mg Capsule; Drug: Placebo oral capsule
- Nemonoxacin 750Mg Capsule (Experimental)
  Interventions: Drug: Nemonoxacin 500Mg Capsule; Drug: Moxifloxacin 400Mg Tablet; Drug: Nemonoxacin 750Mg Capsule; Drug: Placebo oral capsule
- Placebo oral capsule (Placebo Comparator)
  Interventions: Drug: Nemonoxacin 500Mg Capsule; Drug: Moxifloxacin 400Mg Tablet; Drug: Nemonoxacin 750Mg Capsule; Drug: Placebo oral capsule
- Moxifloxacin 400Mg Tablet (Active Comparator)
  Interventions: Drug: Nemonoxacin 500Mg Capsule; Drug: Moxifloxacin 400Mg Tablet; Drug: Nemonoxacin 750Mg Capsule; Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Nemonoxacin 500Mg Capsule — Receive a single dose in a fasting state
  Other Names: TG-873870 500Mg
Drug: Moxifloxacin 400Mg Tablet — Receive a single dose in a fasting state
Drug: Nemonoxacin 750Mg Capsule — Receive a single dose in a fasting state
  Other Names: TG-873870 750Mg
Drug: Placebo oral capsule — Receive a single dose in a fasting state

SUMMARY:
A randomized, single-center, placebo and positive control, 4-period and 4-crossover clinical study with the following main purposes: (1) To evaluate the effect of a single-dose oral administration of nemonoxacin malate capsule on QTc intervals and heart rhythms of healthy subjects. (2) To evaluate the influence of food intake on QTc intervals and pharmacokinetic characteristics.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged between 18 and 40 during the screening period.
2. A volunteer's Body Mass Index (BMI) had to be between 19~24 kg/m2, and a male volunteer's body weight was no less than 50 kg, while female, no less than 45 kg.
3. A subject was judged as a healthy one by investigators according to his/her medical history, physical examination, 12-lead ECG examination, and laboratory test results.
4. A female subject:

   1. was post-menopausal for at least 1 year, or
   2. had been surgically sterilized, or
   3. met the following conditions if she was fertile: (i)her urine pregnancy test results were negative before she started the trial, and (ii)she agreed to use an approved birth control method (e.g. oral contraceptive, spermicide, condom, or intrauterine contraceptive device) throughout the study, and agreed to continue using birth control method within 1 month after the study, and (iii)she may not breastfeed.
5. A male subject had to use a reliable birth control method (using a condom, or his partner executed the foresaid criteria) throughout the study and within 1 month after the study.
6. A subject had never used tobacco or nicotine products within 1 month before receiving the study drug.
7. A subject had never drunk alcohol or drunk more than 12 times within 3 months before receiving the study drug.
8. A subject was willing to completely abstain from foods or beverages containing caffeine or xanthine such as coffee, tea, chocolate, alcohol, grapefruit juice, orange juice, etc within 24 hours before receiving the study drug and during his/her Stage I ward stay.
9. A subject was willing to sign the Informed Consent Form.

Exclusion Criteria:

1. had any personal or family history of sudden cardiac death, myocardial ischemia, myocardial infarction, congestive heart failure, long QT syndrome, hypokalemia, myocarditis, exertional dyspnea, cerebrovascular accident, venous thromboembolism, etc; or
2. needed to use medicine to treat QTc interval prolongation (e.g. Category I or III antiarrhythmic drugs, please refer to Appendix 1) or medicine to treat heart disease; or
3. was found to have abnormal mean values of parameters in 12-lead ECG during the screening: PR >240 ms, QRS >110 ms, male QTcF >430 ms (the automated machine-derived QTcF results in Lead II ECG were used and needed to be confirmed by the investigators), female QTcF >450 ms (the automated machine-derived QTcF results in Lead II ECG were used and needed to be confirmed by the investigators), bradycardia (heart rate <50 bpm); or
4. had clinical abnormalities in 12-lead ECG during screening (e.g. atrioventricular block, torsades de pointes (TdP), other types of ventricular tachycardia, ventricular fibrillation and ventricular flutter, clinically significant T wave changes, or any 12-lead ECG abnormalities that may influence QTc intervals); or
5. had systolic blood pressure >140 mmHg or <90 mmHg, diastolic blood pressure >90 mmHg, pulse <50 bpm or >100 bpm during the screening; or
6. had a positive result in hepatitis B virus or hepatitis C virus serology test; or
7. had a positive pregnancy test result or was currently in lactation period; or
8. was found to have any laboratory test value that was outside the reference value (normal value±10%) during the screening, and that was deemed to have clinical significance by investigators; or
9. had a history of diabetes or cardiovascular disease, liver disease or kidney disease; or
10. had malabsorption syndrome or any other gastrointestinal disease that may influence drug absorption; or
11. had any history of epileptic seizures, or mental disease that may affect protocol compliance, or had a suicidal risk, or had history of alcohol or prohibited drug abuse; or
12. had any disease known to severely affect the immune system, e.g. history of human immunodeficiency virus (HIV) infection, hematologic or solid organ malignancy, or had a splenectomy, etc; or
13. had a hypersensitive idiosyncrasy or hypersensitivity to any drugs, including quinolones or fluoroquinolones; or
14. had a surgery or trauma history within 6 months before receiving the study drug; or
15. had, as shown from his/her medical history, used any known liver enzyme inducer or liver enzyme inhibitor such as benzedrine, barbiturates, benzodiazepines, cannabinoids, cocaine, opiates, phencyclidine, etc within 30 days before receiving the study drug; or
16. had used any other trial drugs within 30 days before receiving the study drug; or
17. had used any prescription drugs or Chinese herbal medicines within 14 days before receiving the study drug; or
18. had used any OTC drugs or nutrition supplements (including the products containing multivalent cation such as calcium, aluminum, magnesium, iron, and zinc, as well as sucralfate, antacids, nutrition supplements, vitamin complex, and dietary metal supplements, etc) within 7 days before receiving the study drug; or
19. had donated ≥400 ml of blood within 3 months before drug administration; or
20. had, as judged by the investigators, any past or current disease or physical condition that may affect the safety or effect evaluation of the study drug; or
21. was identified by the investigators as unsuitable to participate in the study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2012-06-25 (Actual); Primary Completion 2012-08-10 (Actual); Study Completion 2012-08-10 (Actual)

PRIMARY OUTCOMES:
ECG analysis - baseline-adjusted mean QTcF | 2 days
  To compare the post-dosing placebo-corrected, baseline-adjusted mean QTcF differences (ΔΔQTcF) of nemonoxacin 500 mg/750 mg groups and placebo group at corresponding time points with the manually measured QTcF in Lead II of ECG.

SECONDARY OUTCOMES:
ECG analysis - baseline-adjusted mean QTcB | 2 days
  To compare the post-dosing placebo-corrected, baseline-adjusted mean QTcB differences (ΔΔQTcF) of nemonoxacin 500 mg/750 mg groups and placebo group at corresponding time points with the manually measured QTcB in Lead II of ECG.
ECG analysis - baseline-adjusted mean QTcP | 2 days
  To compare the post-dosing placebo-corrected, baseline-adjusted mean QTcP differences (ΔΔQTcF) of nemonoxacin 500 mg/750 mg groups and placebo group at corresponding time points with the manually measured QTcP in Lead II of ECG.
Safety analysis | 33 days
  An analysis of adverse event (number and percentage of subjects) was conducted based on dosage groups
Maximum Plasma Concentration (Cmax) | 2 day
  The analysis was conducted using the well-validated software (WinNolin and DAS programs). A non-compartment model was used to analyze the plasma concentration-time data of nemonoxacin and moxifloxacin, thus the pharmacokinetic parameter was evaluated, and a descriptive summary of the plasma concentration-time data by dosage groups and time points were presented. Also, a descriptive summary of pharmacokinetic parameters were made based on dosage groups.
Time at Which Maximum Plasma Concentration was Observed (Tmax) | 2 day
  The analysis was conducted using the well-validated software (WinNolin and DAS programs). A non-compartment model was used to analyze the plasma concentration-time data of nemonoxacin and moxifloxacin, thus the pharmacokinetic parameter was evaluated, and a descriptive summary of the plasma concentration-time data by dosage groups and time points were presented. Also, a descriptive summary of pharmacokinetic parameters were made based on dosage groups.
Area Under the Plasma Concentration-Time Curve Calculated to the Last Measured Concentration (AUC(0~t)) | 2 day
  The analysis was conducted using the well-validated software (WinNolin and DAS programs). A non-compartment model was used to analyze the plasma concentration-time data of nemonoxacin and moxifloxacin, thus the pharmacokinetic parameter was evaluated, and a descriptive summary of the plasma concentration-time data by dosage groups and time points were presented. Also, a descriptive summary of pharmacokinetic parameters were made based on dosage groups.
Area Under the Plasma Concentration-Time Curve Extrapolated to Infinity (AUC(0~∞)) | 2 day
  The analysis was conducted using the well-validated software (WinNolin and DAS programs). A non-compartment model was used to analyze the plasma concentration-time data of nemonoxacin and moxifloxacin, thus the pharmacokinetic parameter was evaluated, and a descriptive summary of the plasma concentration-time data by dosage groups and time points were presented. Also, a descriptive summary of pharmacokinetic parameters were made based on dosage groups.
Lambda-z (λz) | 2 day
  The analysis was conducted using the well-validated software (WinNolin and DAS programs). A non-compartment model was used to analyze the plasma concentration-time data of nemonoxacin and moxifloxacin, thus the pharmacokinetic parameter was evaluated, and a descriptive summary of the plasma concentration-time data by dosage groups and time points were presented. Also, a descriptive summary of pharmacokinetic parameters were made based on dosage groups.
half-life (t1/2) | 2 day
  The analysis was conducted using the well-validated software (WinNolin and DAS programs). A non-compartment model was used to analyze the plasma concentration-time data of nemonoxacin and moxifloxacin, thus the pharmacokinetic parameter was evaluated, and a descriptive summary of the plasma concentration-time data by dosage groups and time points were presented. Also, a descriptive summary of pharmacokinetic parameters were made based on dosage groups.
Oral Clearance (CLt/F) | 2 day
  The analysis was conducted using the well-validated software (WinNolin and DAS programs). A non-compartment model was used to analyze the plasma concentration-time data of nemonoxacin and moxifloxacin, thus the pharmacokinetic parameter was evaluated, and a descriptive summary of the plasma concentration-time data by dosage groups and time points were presented. Also, a descriptive summary of pharmacokinetic parameters were made based on dosage groups.

REFERENCES:
- [Derived] Zhao C, Lv Y, Li X, Hou F, Ma X, Wei M, Kang Z, Cui L, Xia Y, Liu Y, Tian J. Effects of Nemonoxacin on Thorough ECG QT/QTc Interval: A Randomized, Placebo- and Positive-controlled Crossover Study in Healthy Chinese Adults. Clin Ther. 2018 Jun;40(6):983-992. doi: 10.1016/j.clinthera.2018.04.014. Epub 2018 May 24. PMID 29803534